CLINICAL TRIAL: NCT02217488
Title: Single Ascending Dose Tolerability Study of DG3173
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aspireo Pharmaceuticals Limited (Industry)
Collaborators: DeveloGen AG, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DG3173-I-001
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — PTR 3173

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DG3173 (Experimental)
  Interventions: Drug: DG3173
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DG3173
  Arms: DG3173
Drug: Placebo
  Arms: Vehicle

SUMMARY:
This clinical trial investigated the safety, tolerability and pharmacokinetic profile of DG3173 in a double-blind, randomized, placebo-controlled, single dose escalation Phase 1 study involving 72 healthy volunteers. Individuals received up to 2000 µg of DG3173 via single dose subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic origine: Caucasian
* Weight: 55-95 kg
* BMI: 19-29 kg/qm
* Medical history without clinically relevant pathologies
* Physical examination parameters and lung function without signs of clinically relevant pathologies
* Electrocardiogram recording without signs of clinically relevant pathology, in particular QTc (Bazett) <440ms
* Values for hematology, biochemistry and for coagulation tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the medical investigator (in particular normal values for ALAT, ASAT, LDH, gamma-GT, alkaline phosphatase, alpha-amylase and bilirubin)
* Having given written informed consent before any study-related activities are carried out

Exclusion Criteria:

* Evidence of clinically relevant pathology or disease
* Any history of moderate or severe hypertension, hypotension or orthostatic hypotension
* Mental handicap
* Legal incapacity
* Any history of clinically important emotional and/or psychiatric illness or of any clinically important neurological disorders and/or epilepsy
* Chronic diarrhea or other chronic gastrointestinal disorders
* Acute or chronic gastro-duodenal ulcers
* Presence or history of endocrine disorders
* Presence or history of gall stone disease, presence excluded by means of upper abdominal ultrasound
* Known hypersensitivity to the study drug or constituent of the study drug
* History of any relevant allergy, especially drug and/or food allergies
* Strict vegetarian
* Regular treatment with medications during three months prior to randomization
* Receipt of any prescription or non-prescription medication, including multi-vitamin preparations within 14 days prior to drug administration and for the duration of the study
* Use of St. John´s Wort or Ginkgo Biloba (also known as Ginkgo Bilbao) within 48 hours prior to randomization
* Participation in a clinical study within 30 days prior to randomization
* Donation of blood within 60 days prior to randomization
* History of use of tobacco or nicotine-containing products within the past three months
* Any history of alcohol abuse or drug addiction
* Positive results at screen for drugs of abuse (cocaine, amphetamine/methamphetamine, tetrahydrocannbinol, opiates) or alcohol (breath test) at screening or on admission
* Positive screen results for HBsAg, anti-HCV, or anti-HIV1&2
* Consumption of abnormal quantities of coffee or tea (i.e. more than 5 cups per day [1 cup = 150 ml]
* Any disease which in the Investigator´s opinion would exclude the subject from the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events or withdrawals due to adverse events | One week